CLINICAL TRIAL: NCT02610933
Title: The Effect of Replacement of Vitamin K Antagonist by Rivaroxaban With or Without Vitamin K2 Supplementation on Vascular Calcifications in Chronic Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Effect on Vascular Calcification of Replacing Warfarin by Rivaroxaban With or Without VitK2 in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Rogier Caluwe, Dr. Rogier Caluwé, MD, Onze Lieve Vrouw Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014/065
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Vascular Calcification
Keywords: vascular calcification; hemodialysis; rivaroxaban; vitamin K2
MeSH Terms: conditions — Vascular Calcification | interventions — Rivaroxaban; Vitamin K 2

ARMS (3):
- Vitamin K antagonist (No Intervention): Vitamin K antagonist treatment targeting an international normalized ratio of 2 to 3 for 18 months
- rivaroxaban (Active Comparator): Rivaroxaban 10 mg tablet by mouth once daily for 18 months
  Interventions: Drug: rivaroxaban
- rivaroxaban and vitamin K2 (Active Comparator): Rivaroxaban 10 mg tablet by mouth once daily and MK-7 2000 microgram tablet by mouth thrice weekly for 18 months
  Interventions: Drug: rivaroxaban; Dietary Supplement: Vitamin K2

INTERVENTIONS:
Drug: rivaroxaban — replacement of vitamin K antagonist by rivaroxaban
  Arms: rivaroxaban; rivaroxaban and vitamin K2
Dietary Supplement: Vitamin K2 — Vitamin K2 supplementation
  Other Names: MK-7
  Arms: rivaroxaban and vitamin K2

SUMMARY:
This study examines patients on chronic hemodialysis with non-valvular atrial fibrillation, who have a CHA2DS2-VASc Score of ≥ 2 and therefore are candidates for or already receive a vitamin K antagonist.

The first question is whether replacement of the vitamin K antagonist by rivaroxaban is able to slow progression of vascular calcification. The second question is whether addition of vitamin K2 to rivaroxaban can further slow down or even halt the progression of vascular calcification.

DETAILED DESCRIPTION:
The present study targets dialysis patients with non-valvular atrial fibrillation requiring treatment with vitamin K antagonists. It addresses the question whether replacement of the vitamin K antagonist by rivaroxaban is able to slow progression of vascular calcification (VC). The second research question is whether addition of vitamin K2 to rivaroxaban can further beneficially affect the progression of VC. Two non-invasive methods are used to evaluate the impact of interventions on the progression of VC: i.e. coronary artery calcification (CAC) and pulse wave velocity (PWV) measurements. The detection of CAC is predictive for the presence of obstructive coronary artery disease and future coronary events. VC and stiffening of the central elastic-type arteries are independent predictors of cardiovascular morbidity and mortality in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* end stage renal failure treated with chronic hemodialysis
* atrial fibrillation
* CHA2DS2-VASc Score ≥ 2
* ability to provide informed consent

Exclusion Criteria:

* known intestinal malabsorption or inability to take oral medication
* inability to stop co-medication that causes major interactions with rivaroxaban (e.g. ketoconazole, itraconazole, voriconazole, posaconazole, ritonavir, rifampicin, phenytoin, carbamazepine, phenobarbital or St John's wort)
* investigator's assessment that the subject's life expectancy is less than 1 year
* prosthetic mechanical heart valve
* contraindication for anticoagulation
* liver dysfunction Child-Pugh grade B-C
* pregnancy, breastfeeding, inadequate contraception
* incompliance with medication and scheduled investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-11; Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
absolute and relative change in coronary artery calcification score | 18 months
  score measured by unenhanced electrocardiographically-gated CT of the heart and thoracic aorta and calculated on 2.5 mm slices using Smartscore v.4.0 (GE Healthcare)
absolute and relative change in thoracic aortic calcification score | 18 months
  score measured by unenhanced electrocardiographically-gated CT of the heart and thoracic aorta and calculated on 2.5 mm slices using Smartscore v.4.0 (GE Healthcare)
absolute and relative change in pulse wave velocity | 18 months

SECONDARY OUTCOMES:
absolute and relative change in aortic valve calcification score | 18 months
  score measured by unenhanced electrocardiographically-gated CT of the heart and thoracic aorta and calculated on 2.5 mm slices using Smartscore v.4.0 (GE Healthcare)
absolute and relative change in mitral valve calcification score | 18 months
  score measured by unenhanced electrocardiographically-gated CT of the heart and thoracic aorta and calculated on 2.5 mm slices using Smartscore v.4.0 (GE Healthcare)
mortality from any cause | 18 months
myocardial infarction, acute coronary syndrome, symptom-driven coronary revascularization and death from cardiovascular cause | 18 months
Stroke, defined as sudden onset of focal neurological deficit consistent with the territory of a major cerebral artery and categorised as ischaemic, haemorrhagic, or unspecified. | 18 months
Systemic embolism, defined as an acute vascular occlusion of a limb or organ documented by imaging, surgery, or autopsy. | 18 months
Major bleeding, defined as a requirement for transfusion of two or more units of blood or a decrease in haemoglobin of 2 g/dL or more. | 18 months
Life-threatening bleeding, defined as fatal bleeding, symptomatic intracranial bleeding, a decrease in haemoglobin of 5 g/dL or more, or a requirement for transfusion of four or more units of blood, inotropic agents, or surgery. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Rogier Caluwé, MD, Principal Investigator — Nephrology Department OLV Hospital Aalst Belgium
Locations (1):
- OLV Hospital, Aalst, Belgium

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593